CLINICAL TRIAL: NCT07123909
Title: The Use of Sorption Technologies in Patients Receiving Program Hemodialysis With Inflammatory Syndrome
Brief Title: Studies on Adsorption International Learning Initiative Global
Acronym: SAILING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Botkin Hospital (Other)
Responsible Party: Principal Investigator, Evgeny Shutov, Head of the Nephrology Center, Botkin Hospital, Botkin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-4/27012025
Record Dates: First submitted 2025-07-04; First posted 2025-08-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D; Uremia; Chronic; Uremic; Toxemia; Inflammation Chronic; Hemodialysis; Inflammation Biomarkers; Dialysis Related Complication; Anemia Associated With End Stage Renal Disease
Keywords: Program dialysis; Sorption; Complications of program dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia; Bronchiolitis Obliterans Syndrome; Toxemia | interventions — Hemoperfusion; Sorption Detoxification

STUDY DESIGN:
Intervention Model Description: This study will comprise two groups of 30 participants each. The intervention group will receive standard hemodialysis with adjunctive hemosorption therapy using the Jafron HA130 cartridge, while the control group will receive standard hemodialysis treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of hemodialysis and hemosorption (Experimental): Dialysis patients will undergo a combined procedure of hemodialysis and hemosorption using the Jafron HA130 cartridge three times per week during the first month, twice per week in the second month, and once per week in the third month.
  Interventions: Device: Patients will undergo a combined hemodialysis and hemosorption procedure. The study cartridge for hemosorption by Jafron HA130 contains the original adsorbing material.
- Standard hemodialysis procedure (No Intervention): Dialysis patients on standard dialysis procedure

INTERVENTIONS:
Device: Patients will undergo a combined hemodialysis and hemosorption procedure. The study cartridge for hemosorption by Jafron HA130 contains the original adsorbing material. — The test cartridge will be used in addition to the ongoing program hemodialysis three times a week in the first month, twice a week in the next month, once a week in the third month
  Other Names: Jafron HA130; hemosorption; cartridge for hemosorption; Sorption; Program dialysis
  Arms: Combination of hemodialysis and hemosorption

SUMMARY:
Use of sorption technologies in patients undergoing maintenance hemodialysis with inflammatory syndrome and clinical manifestations of uremia

DETAILED DESCRIPTION:
This study will involve 30 hemodialysis patients selected based on examination results showing elevated C-reactive protein (CRP) and/or interleukin-6 (IL-6) levels. Participants will undergo hemoadsorption with the Jafron HA130 cartridge performed concurrently with hemodialysis: three times per week during the first month, twice per week during the second month, and once per week during the third month.

The following parameters will be assessed: inflammatory markers (CRP, IL-1, IL-6, IL-8, β2-microglobulin, free light chains of immunoglobulins), parathyroid hormone (PTH), standard biochemical blood tests (creatinine, urea, calcium, phosphorus, albumin, iron metabolism), and complete blood count. Analyses will be performed at baseline (before inclusion) and monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate dialysis defined by a KT/V index ≥ 1.4
2. No active inflammatory process or infection
3. Age ≥ 18 years
4. Receiving standard hemodialysis regimen three times weekly, at least 4 hours per session
5. Participants with elevated interleukin-6 (IL-6) and/or C-reactive protein (CRP) levels exceeding local laboratory reference values

Exclusion Criteria:

1. Current use of steroids or immunosuppressive therapy
2. History of kidney transplantation
3. Diagnosis of cancer
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum IL-6, pg/ml | By the third month

SECONDARY OUTCOMES:
Change frome baseline in serum IL-1, pg/ml | Monthly for 3 months
Change from baseline in serum IL-8, pg/ml | Monthly for 3 months
Change from baseline in serum IL-10, pg/ml | Monthly for 3 months
Change from baseline in CRP, mg/L | Monthly for 3 months
Change from baseline in β2-microglobulin, mg/L | Monthly for 3 months
Change from baseline in free light chains, mcg/ml | Monthly for 3 months
Change from baseline in PTH, pg/ml | Monthly for 3 months
Change from baseline in serum iron, mcg/dL | Monthly for 3 months
Change from baseline in ferritin, mcg/L | Monthly for 3 months
Change from baseline in saturated transferrin, TS% | Monthly for 3 months
Change from baseline in albumin, g/L | Monthly for 3 months
Change from baseline in phosphorus, mmol/L | Monthly for 3 months
Change from baseline in calcium, mmol/L | Monthly for 3 months
Change from baseline in blood urea nitrogen (BUN), mmol/L | Monthly for 3 months
Change from baseline in creatinine, mg/dL | Monthly for 3 months
Change from baseline in hemoglobin (Hb), g/L | Monthly for 3 months
Change from baseline in Hospital Anxiety and Depression Scale Score | Monthly for 3 months
  Scale consists of two subscales. The minimum score of each is 0, and the maximum score on each of the two subscales is 21. The higher the score, the higher the level of anxiety and depression.
Change from baseline in pruritus (Visual Analogue Scale) | Monthly for 3 months
  From 0 to 10 where 10 is maximum

CONTACTS AND LOCATIONS:
Locations (1):
- Botkin Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT07123909/Prot_000.pdf